CLINICAL TRIAL: NCT00899028
Title: Identification and Validation of Molecular Markers in Lung Cancer
Brief Title: Identifying Biomarkers for Lung Cancer Using Tissue Samples From Patients With Lung Cancer and From Healthy Participants
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pierre P. Massion, Professor, Vanderbilt University Medical Center
Other Study IDs: CDR0000584223; R01CA102353 (NIH); P30CA068485 (NIH); VU-VICC-THO-0373; VU-VICC-010178
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: stage 0 non-small cell lung cancer; stage I non-small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer; stage II non-small cell lung cancer; stage IV non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Comparative Genomic Hybridization; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: comparative genomic hybridization
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry
Other: medical chart review
Procedure: diagnostic bronchoscopy

SUMMARY:
RATIONALE: Studying samples of tissue, blood, sputum, and urine from patients with lung cancer and from healthy participants in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers for lung cancer using tissue samples from patients with lung cancer and from healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify new molecular abnormalities specific to the development of squamous cell carcinoma of the lung.
* To determine the prevalence of candidate biomarkers in lung cancer progression.
* To determine the odds of developing lung cancer according to biomarker status in preinvasive lesions.
* To determine the odds of developing lung cancer according to proteomic biomarker status in the normal bronchial epithelium of high-risk patients.

OUTLINE: This is a multicenter study.

Tissue samples are collected at the time of fluorescence bronchoscopy for laboratory biomarker studies. Blood, sputum, and urine samples are also collected. Gene and protein expression studies are performed on the samples using comparative genomic hybridization array, 3q oligonucleotide microarray, matrix-assisted laser desorption/ionization time of flight mass spectrometry (MALDI-TOF), fluorescence in situ hybridization (FISH), and immunohistochemistry (IHC).

Patients' medical records are reviewed to collect information about the patient's past medical history and pertinent laboratory and radiography results.

Patients and healthy volunteers are followed annually via telephone or a mailed questionnaire.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Known or previously diagnosed lung cancer
  * Suspected lung cancer, including the following:

    * Completely resected stage I lung cancer (with no evidence of metastatic disease) for which patient is at risk for developing secondary disease
    * Suspected of having lung cancer due to clinical symptoms, such as positive sputum cytology, hemoptysis, unresolved pneumonia, persistent cough, and positive x-ray
  * Healthy volunteer

PATIENT CHARACTERISTICS:

* WBC ≥ 2,000/mm³ but ≤ 20,000/mm³
* Platelet count ≥ 50,000/mm³
* Not pregnant
* No uncontrolled hypertension (i.e., systolic blood pressure > 200 mm Hg, diastolic blood pressure > 120 mm Hg)
* No unstable angina
* No known bleeding disorder
* No other contraindications for white light bronchoscopic examination
* No other contraindications for fluorescence examination

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior fluorescent photosensitizing agents (hematoporphyrin derivatives)
* More than 3 months since prior and no concurrent chemopreventative drugs (e.g., tretinoin)
* More than 6 months since prior ionizing radiation treatment to the chest
* More than 6 months since prior systemic cytotoxic chemotherapy
* No concurrent anticoagulant therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2001-05; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Identification of new molecular markers specific to the development of squamous cell lung cancer
Prevalence of candidate biomarkers in lung cancer progression
Odds of developing lung cancer according to biomarker status

CONTACTS AND LOCATIONS:
Overall Officials: Pierre P. Massion, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee